CLINICAL TRIAL: NCT00179972
Title: Evaluation of Pulse Oximetry Sensors in Neonates
Status: Terminated | Type: Observational
Why Stopped: Lack of resources and loss of personnel precluded study progress. No adverse events or unanticipated problems involving risks to subjects.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2005-196N
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Premature Birth
Keywords: Pulse oximetry; Pulse oximetry sensors; Skin Integrity; Prematurity; Neonatal Intensive Care Unit; Infant, premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Adhesive and non-adhesive oximetry sensors — A sample of 32 premature infants will be recruited to participate in this study in which an adhesive sensor and a nonadhesive sensor are compared. Both sensors will be simultaneously tested in each subject, for a period of 14 days, with one sensor on the right foot and the other sensor on the left foot. Data will be collected on sensor longevity, skin integrity at the sensor site, reason for sensor replacement and ease of use rating by the clinician. Data will be summarized using descriptive statistics.

SUMMARY:
The purpose of this study is to evaluate sensor longevity and skin integrity with two different models of neonatal pulse oximetry sensors currently used for monitoring oxygen levels in small infants.

DETAILED DESCRIPTION:
A common method for assessing the respiratory status of hospitalized children is the use of pulse oximetry. This noninvasive device typically is placed on a finger, foot/palm of a child. Red and infrared light is shined through the tissue under the sensor and the information is sent back to a monitor for calculation of oxygen saturation. Use of this noninvasive method provides continuous information on the oxygenation status of patients and has greatly reduced the number of arterial blood samples required for patient care.

While the advantages of noninvasive pulse oximetry are significant, there are a number of factors which can negatively impact the performance of the device. Patient movement and sensor adherence to the skin have been some of the challenges to optimal device performance. While much of the clinical research on pulse oximetry sensors over the years has evaluated device accuracy and reliability, limited data is available on sensor longevity under conditions typical of clinical use. A particular challenge with neonatal pulse oximetry monitoring is insuring proper sensor adherence within the warm, moist environment of incubators used in neonatal care. Furthermore, limited data are available on the impact of sensor adherence on skin integrity in premature infants who are at high risk for skin breakdown.

Objectives. The purpose of this study is to evaluate sensor longevity and impact on skin integrity in neonatal patients with two different models of pulse oximetry sensors.

Research Method. A sample of 32 premature infants will be recruited to participate in this study in which an adhesive sensor and a nonadhesive sensor are compared. Both sensors will be simultaneously tested in each subject, for a period of 14 days, with one sensor on the right foot and the other sensor on the left foot. Data will be collected on sensor longevity, skin integrity at the sensor site, reason for sensor replacement and ease of use rating by the clinician. Data will be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 34 weeks
* Weight < 3.0 kg
* Postnatal age < 2 weeks
* Anticipated pulse oximetry monitoring for at least 14 days

Exclusion Criteria:

* Presence of any skin irritation or breakdown on either foot
* Foot impediments which would preclude proper placement of the test sensors
* Known allergies to adhesive materials

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: NICU of Ann & RObert H. Lurie Children's Hospital of CHicago
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2005-09; Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Fleming, RNC, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States